CLINICAL TRIAL: NCT07248345
Title: A Machine Learning-enhanced Virtual Reality Intervention to Facilitate Balance Finding for Family Caregivers of Persons Living With Dementia
Brief Title: Virtual Reality Intervention for Family Caregivers of Persons Living With Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 114-2314-B-182-048-MY3
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Dementia
Keywords: family caregiver; dementia; virtual reality
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality (Experimental): virtual interventions using VR scenarios related to competing demands for family caregivers of PLWD
  Interventions: Behavioral: virtual reality intervention
- information (No Intervention): information regarding dementia will be provided

INTERVENTIONS:
Behavioral: virtual reality intervention — virtual interventions using VR scenarios related to competing demands for family caregivers of PLWD
  Arms: virtual reality

SUMMARY:
This study explores the effects of a virtual reality intervention on family caregivers of persons living with dementia

DETAILED DESCRIPTION:
Virtual interventions using VR scenarios related to competing demands for family caregivers of persons living with dementia that facilitate caregiving balance will be developed. Tts effects will be investigated by using a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

- has the primary responsibility for providing direct care or supervising the care received by the PLWD, and is living with the PLWD.

Exclusion Criteria:

-

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Caregiving Balance | 1st month follwing VR intervention
  The balance between competing needs will be assessed using the Caregiving Process of Finding a Balance Point scale
Caregiving Balance | 3rd month follwing VR intervention
  The balance between competing needs will be assessed using the Caregiving Process of Finding a Balance Point scale
Caregiving Balance | 6th month follwing VR intervention
  The balance between competing needs will be assessed using the Caregiving Process of Finding a Balance Point scale
Caregiver role strain | 1st month following VR intervention
  Role strain will be measured by the 87-item Role Strain Scale from the Family Caregiving Inventory (FCI)
Caregiver role strain | 3rd month following VR intervention
  Role strain will be measured by the 87-item Role Strain Scale from the Family Caregiving Inventory (FCI)
Caregiver role strain | 6th month following VR intervention
  Role strain will be measured by the 87-item Role Strain Scale from the Family Caregiving Inventory (FCI)

SECONDARY OUTCOMES:
Health Related Quality of Life | 1st month following VR intervention
  Physical functioning, role physical, bodily pain, vitality, general health, social functioning, role emotional, and mental health will be assessed with the 36-item Short Form Health Survey (SF-36 ).
Health Related Quality of Life | 3rd month following VR intervention
  Physical functioning, role physical, bodily pain, vitality, general health, social functioning, role emotional, and mental health will be assessed with the 36-item Short Form Health Survey (SF-36 ).
Health Related Quality of Life | 6th month following VR intervention
  Physical functioning, role physical, bodily pain, vitality, general health, social functioning, role emotional, and mental health will be assessed with the 36-item Short Form Health Survey (SF-36 ).
Depressive symptoms | 1st month following VR intervention
  The Chinese version of the 20-item Center for Epidemiologic Studies Depression Scale (CES-D will assess depressive symptoms.
Depressive symptoms | 3rd month following VR intervention
  The Chinese version of the 20-item Center for Epidemiologic Studies Depression Scale (CES-D will assess depressive symptoms.
Depressive symptoms | 6th month following VR intervention
  The Chinese version of the 20-item Center for Epidemiologic Studies Depression Scale (CES-D will assess depressive symptoms.
Caregiving Rewards | 1st month following VR intervention
  The FCI Rewards of Caregiving scale (Archbold, et al., 1990) will be used to assess positive outcomes of caregiving
Caregiving Rewards | 3rd month following VR intervention
  The FCI Rewards of Caregiving scale (Archbold, et al., 1990) will be used to assess positive outcomes of caregiving
Caregiving Rewards | 6th month following VR intervention
  The FCI Rewards of Caregiving scale (Archbold, et al., 1990) will be used to assess positive outcomes of caregiving

OTHER OUTCOMES:
Caregiving demands | 1st month following VR intervention
  The FCI Caregiving Activities Scales (Archbold, et al., 1990) will measure caregiving demand.
Caregiving demands | 3rd month following VR intervention
  The FCI Caregiving Activities Scales (Archbold, et al., 1990) will measure caregiving demand.
Caregiving demands | 6th month following VR intervention
  The FCI Caregiving Activities Scales (Archbold, et al., 1990) will measure caregiving demand.

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Ing Shyu, Principal Investigator — Chang Gung University

IPD SHARING:
Plan to Share IPD: No